CLINICAL TRIAL: NCT01993719
Title: A Phase II Study for Metastatic Melanoma Using High-Dose Chemotherapy Preparative Regimen Followed by Cell Transfer Therapy Using Tumor-Infiltrating Lymphocytes Plus IL-2 With the Administration of Pembrolizumab in the Retreatment Arm
Brief Title: Immunotherapy Using Tumor Infiltrating Lymphocytes for Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Stephanie Goff, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 140022; 14-C-0022
Record Dates: First submitted 2013-11-22; First posted 2013-11-25 (Estimated); Results first posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-12

CONDITIONS: Metastatic Melanoma
Keywords: Melanoma; Adoptive Cell Therapy
MeSH Terms: conditions — Melanoma | interventions — aldesleukin; fludarabine; fludarabine phosphate; Cyclophosphamide; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm 1N -Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin (Experimental): Standard Chemo Prep Regimen. Young Tumor Infiltrating Lymphocytes (TIL) Plus High Dose Interleukin-2, Standard Chemo Preparative Regimen in participants without prior treatment pembrolizumab or nivolumab Standard preparative regimen + Young Tumor Infiltrating Lymphocytes (TIL) Cells Aldesleukin: 720,000 IU/kg intravenous (IV) every eight hours (+/- 1 hour) beginning within 24 hours of cell infusion and continuing for up to 4 days (maximum 12 doses).
  Fludarabine: 25 mg/m^2/day intravenous piggy-back (IVPB) daily for 5 days Cyclophosphamide: 60 mg/kg/day X 2 days intravenous (IV) Young TIL: Day 0: Cells will be infused intravenously (IV)
  Interventions: Drug: Aldesleukin; Drug: Fludarabine; Drug: Cyclophosphamide; Biological: Young TIL
- Arm 1P - Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin (Experimental): Standard Chemo Prep Regimen Young Tumor Infiltrating Lymphocytes (TIL) Plus High Dose Interleukin-2, Standard Chemo Preparative Regimen in participants previously treated with pembrolizumab or nivolumab.
  Standard preparative regimen + Young Tumor Infiltrating Lymphocytes (TIL) Cells Aldesleukin: 720,000 IU/kg intravenous (IV) every eight hours (+/- 1 hour) beginning within 24 hours of cell infusion and continuing for up to 4 days (maximum 12 doses).
  Fludarabine: 25 mg/m^2/day intravenous piggy-back (IVPB) daily for 5 days Cyclophosphamide: 60 mg/kg/day X 2 days intravenous (IV) Young TIL: Day 0: Cells will be infused intravenously (IV)
  Interventions: Drug: Aldesleukin; Drug: Fludarabine; Drug: Cyclophosphamide; Biological: Young TIL
- Arm 2/Foll By Arm 1P-Low dose Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin (Experimental): Decreased Chemo Prep Regimen+Retreat. Young TIL+High Dose Interleukin-2, Decreased Chemo Preparative Regimen. Young TIL+High Dose Interleukin-2, Standard Chemo (Retreat). Lower dose preparative regimen + Young TIL Cells. Aldesleukin: 720,000 IU/kg IV every eight hours (+/- 1 hour) beginning within 24 hours of cell infusion and continuing for up to 4 days (maximum 12 doses). Fludarabine: 30 mg/kg/day intravenous piggy-back (IVPB) daily for 3 days. Cyclophosphamide: Days -5 to -3 (low-dose arm): Cyclophosphamide 300 mg/m^2 IV over 60 minutes. Young TIL: Day 0: Cells will be infused IV. Retreatment: Standard Chemo Prep Regimen. Aldesleukin: 720,000 IU/kg IV every eight hours (+/- 1 hour) beginning within 24 hours of cell infusion and continuing for up to 4 days (maximum 12 doses). Fludarabine: 25 mg/m^2/day intravenous piggy-back (IVPB) daily for 5 days. Cyclophosphamide: 60 mg/kg/day X 2 days IV. Young TIL: Day 0: Cells will be infused IV.
  Interventions: Drug: Aldesleukin; Drug: Fludarabine; Drug: Cyclophosphamide; Biological: Young TIL
- Arm 2- Low Dose Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin (Experimental): Decreased Chemo Prep Regimen. Young Tumor Infiltrating Lymphocytes (TIL) Plus High Dose Interleukin-2 Lower Dose preparative regimen + Young Tumor Infiltrating Lymphocytes (TIL) Cells Aldesleukin: 720,000 IU/kg intravenous (IV) every eight hours (+/- 1 hour) beginning within 24 hours of cell infusion and continuing for up to 4 days (maximum 12 doses).
  Fludarabine: 30 mg/kg/day intravenous piggy-back (IVPB) daily for 3 days Cyclophosphamide: Days -5 to -3 (low-dose arm): Cyclophosphamide 30 mg/kg IV over 60 minutes for 2 days.
  Young TIL: Day 0: Cells will be infused intravenously (IV)
  Interventions: Drug: Aldesleukin; Drug: Fludarabine; Drug: Cyclophosphamide; Biological: Young TIL
- Arm 1P/Foll By Arm-1P/R-Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin (Experimental): Standard Chemo Prep Regimen(SCPR)+Retreat. Young TIL+High Dose(HD) Interleukin-2, SCPR. Young TIL+HD Interleukin-2, SC(Retreat). SCPR+Young TIL Cells retreatment with SCPR+Young TIL Cells+pembrolizumab. Aldesleukin:720,000 IU/kgIV every eight hours (+/-1 hour) beginning within 24 hours of cell infusion and continuing for up to 4 days (maximum 12 doses). Fludarabine:25 mg/m^2/day intravenous piggy-back(IVPB) daily for 5 days. Cyclophosphamide:60 mg/kg/day X 2 days IV. Young TIL:Day 0: Cells will be infused IV. Retreatment with standard preparative regimen+Young TIL Cells+pembrolizumab. Aldesleukin:720,000 IU/kg IV every eight hours (+/- 1 hour) beginning within 24 hours of cell infusion and continuing for up to 4 days (maximum 12 doses). Fludarabine:25 mg/m^2/day intravenous piggy-back (IVPB) daily for 5 days. Cyclophosphamide:60 mg/kg/day X 2 days IV. Young TIL: Day 0:Cells will be infused IV. Pembrolizumab:2 mg/kg IV on Days -2, 21 (+/- 2 days), 42 (+/- 2 days), and 63 (+/- 2 days).
  Interventions: Drug: Aldesleukin; Drug: Fludarabine; Drug: Cyclophosphamide; Biological: Young TIL; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Aldesleukin — 720,000 IU/kg intravenous (IV) every eight hours (+/- 1 hour) beginning within 24 hours of cell infusion and continuing for up to 4 days (maximum 12 doses).
  Other Names: Proleukin
Drug: Fludarabine — 25 mg/m^2/day intravenous piggy-back (IVPB) daily for 5 days
  Other Names: Fludara
  Arms: Arm 1N -Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin; Arm 1P - Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin; Arm 1P/Foll By Arm-1P/R-Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin; Arm 2/Foll By Arm 1P-Low dose Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin
Drug: Fludarabine — 30 mg/kg/day intravenous piggy-back (IVPB) daily for 3 days.
  Other Names: Fludara
  Arms: Arm 2- Low Dose Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin; Arm 2/Foll By Arm 1P-Low dose Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin
Drug: Cyclophosphamide — 60 mg/kg/day X 2 days intravenous (IV)
  Other Names: Cytoxan
  Arms: Arm 1N -Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin; Arm 1P - Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin; Arm 1P/Foll By Arm-1P/R-Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin; Arm 2/Foll By Arm 1P-Low dose Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin
Drug: Cyclophosphamide — Days -5 to -3 (low-dose arm):30 mg/kg IV over 60 minutes for 2 days
  Other Names: Cytoxan
  Arms: Arm 2- Low Dose Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin
Drug: Cyclophosphamide — Days -5 to -3 (low-dose arm): 300 mg/m^2 IV over 60 minutes.
  Other Names: Cytoxan
  Arms: Arm 2/Foll By Arm 1P-Low dose Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin
Biological: Young TIL — Day 0: Cells will be infused intravenously (IV)
  Other Names: Young Tumor Infiltrating Lymphocytes
Drug: Pembrolizumab — 2 mg/kg intravenous (IV) on Days -2, 21 (+/- 2 days), 42 (+/- 2 days), and 63 (+/- 2 days).
  Other Names: Keytruda
  Arms: Arm 1P/Foll By Arm-1P/R-Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin

SUMMARY:
Background:

* The National Cancer Institute (NCI) Surgery Branch has developed an experimental therapy that involves taking white blood cells from patients' tumors, growing them in the laboratory in large numbers, and then giving the cells back to the patient. These cells are called Tumor Infiltrating Lymphocytes, or TIL and we have given this type of treatment to over 400 patients with melanoma.
* In this trial, we are determining if there is a difference in the response between patients who have received prior anti-programmed cell death-1 (PD-1) treatment to those who have not received this prior ant-PD1 treatment.

Objectives:

- To determine if there is a difference in the rate of response between patients who have received prior anti-PD1 and those who have not.

Eligibility:

- Individuals at least 18 years and less than or equal to 70 years of age who have metastatic melanoma.

Design:

* Work up stage: Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected.
* Surgery: Surgery or biopsy will be performed to obtain tumor from which to grow white blood cells. White blood cells will be grown from the tumor in the laboratory.
* Leukapheresis: Participants will have leukapheresis to collect additional white blood cells. (Leukapheresis is a common procedure which removes only the white blood cells from the patient.)
* Treatment: Participants will receive standard dose chemotherapy to prepare their immune system to accept the white blood cells. Participants will receive an infusion of their own white blood cells grown from tumor. They will also receive aldesleukin for up to five days to boost the immune system s response to the white blood cells. They will stay in the hospital for about 4 weeks for the treatment.
* Follow up: Patients will return to the clinic for a physical exam, review of side effects, lab tests, and scans about every 1-3 months for the first year, and then every 6 months to 1 year as long as their tumors are shrinking. Follow up visits take up to 2 days.

DETAILED DESCRIPTION:
Background:

* Adoptive cell therapy (ACT) using autologous tumor infiltrating lymphocytes can mediate the regression of bulky metastatic melanoma when administered along with high-dose aldesleukin (IL-2) following a non-myeloablative lymphodepleting chemotherapy preparative regimen consisting of cyclophosphamide and fludarabine.
* In a series of consecutive trials using this chemotherapy preparative regimen alone or with 2 Gray (Gy) or 12 Gy total body irradiation (TBI) objective response rates using Response Evaluation Criteria In Solid Tumors (RECIST) criteria were 49%, 52%, and 72%, respectively. Of the 20 complete regressions seen in this trial, 19 are on-going at 70 to 114 months.
* The chemotherapy alone preparative regimen required in-patient treatment and was associated with significant neutropenia and thrombocytopenia requiring multiple transfusions and treatment for febrile neutropenia.

Objectives:

* With amendment D, to determine if there is a difference in the rate of response between patients who have received prior anti-PD1 and those who have not; both groups will receive non-myeloablative lymphoid depleting preparative regimen followed by autologous young tumor infiltrating lymphocytes (TIL) and administration of high dose aldesleukin.
* To determine the toxicity of the treatment.

Eligibility:

* Age greater than or equal to 18 and less than or equal to 70 years
* Evaluable metastatic melanoma
* Metastatic melanoma lesion suitable for surgical resection for the preparation of TIL
* No contraindications to high-dose aldesleukin administration
* No concurrent major medical illnesses or any form of immunodeficiency

Design:

* Patients with metastatic melanoma will have lesions resected and after TIL growth is established, patients will receive ACT with TIL plus aldesleukin following high dose chemotherapy preparative regimen.
* Up to 64 patients may be enrolled over 4-5 years.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Measurable metastatic melanoma with at least one lesion that is resectable for tumor infiltrating lymphocytes (TIL) generation and at least one other lesion that can be measured by Response Evaluation Criteria In Solid Tumors (RECIST) criteria.
2. Confirmation of diagnosis of metastatic melanoma by the Laboratory of Pathology of National Cancer Institute (NCI).
3. Patients with 3 or fewer brain metastases that are less than 1 cm in diameter and asymptomatic are eligible. Lesions that have been treated with stereotactic radiosurgery must be clinically stable for 1 month after treatment for the patient to be eligible. Patients with surgically resected brain metastases are eligible.
4. Greater than or equal to 18 years of age and less than or equal to 70 years of age.
5. Ability of subject to understand and the willingness to sign the Informed Consent Document
6. Willing to sign a durable power of attorney.
7. Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0, 1 or 2.
8. Patients of both genders must be willing to practice birth control from the time of enrollment on this study and for up to four months after treatment.
9. Serology:

   * Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune-competence and thus are less responsive to the experimental treatment and more susceptible to its toxicities.)
   * Seronegative for hepatitis B antigen, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by reverse transcription polymerase chain reaction (RT-PCR) and be hepatitis C virus (HCV) ribonucleic acid (RNA) negative.
10. Women of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the treatment on the fetus.
11. Hematology:

    * Absolute neutrophil count greater than 1000/mm(3) without the support of filgrastim
    * White blood cell (WBC) greater than or equal to 3000/mm(3)
    * Platelet count greater than or equal to 100,000/mm(3)
    * Hemoglobin > 8.0 g/dl
12. Chemistry:

    * Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less than or equal to 2.5 times the upper limit of normal
    * Serum Creatinine less than or equal to 1.6 mg/dl
    * Total bilirubin less than or equal to 1.5 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.
13. More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patients toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo). Patients must have progressive disease after prior treatment.

    Note: Patients may have undergone minor surgical procedures within the past 3 weeks, as long as all toxicities have recovered to grade 1 or less.
14. Subjects must be co-enrolled in 03-C-0277

EXCLUSION CRITERIA:

1. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the treatment on the fetus or infant.
2. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
3. Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
4. Active systemic infections, (e.g.: requiring anti-infective treatment), coagulation disorders or any other active major medical illnesses.
5. Concurrent systemic steroid therapy.
6. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
7. History of coronary revascularization or ischemic symptoms.
8. Any patient known to have an left ventricular ejection fraction (LVEF) less than or equal to 45%
9. Documented LVEF of less than or equal to 45%, note: testing is required in patients with:

   * Age greater than or equal to 65 years old
   * Clinically significant atrial and or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second or third degree heart block or history of ischemic heart disease or chest pain.
10. Patients who are receiving other investigational agents
11. Documented forced expiratory volume (FEV1) less than or equal to 60% predicted tested in patients with:

    * A prolonged history of cigarette smoking (20 pack (pk)/year of smoking within the past 2 years).
    * Symptoms of respiratory dysfunction

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-12-12 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2022-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie L Goff, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the Study Principal Investigator (PI).

REFERENCES:
- [Background] Dudley ME, Yang JC, Sherry R, Hughes MS, Royal R, Kammula U, Robbins PF, Huang J, Citrin DE, Leitman SF, Wunderlich J, Restifo NP, Thomasian A, Downey SG, Smith FO, Klapper J, Morton K, Laurencot C, White DE, Rosenberg SA. Adoptive cell therapy for patients with metastatic melanoma: evaluation of intensive myeloablative chemoradiation preparative regimens. J Clin Oncol. 2008 Nov 10;26(32):5233-9. doi: 10.1200/JCO.2008.16.5449. Epub 2008 Sep 22. PMID 18809613
- [Background] O'Brien SM, Kantarjian HM, Cortes J, Beran M, Koller CA, Giles FJ, Lerner S, Keating M. Results of the fludarabine and cyclophosphamide combination regimen in chronic lymphocytic leukemia. J Clin Oncol. 2001 Mar 1;19(5):1414-20. doi: 10.1200/JCO.2001.19.5.1414. PMID 11230486
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-C-0022.html

RESULTS

PARTICIPANT FLOW:
Period: First Drug Administration
Arm/Group | Arm 1N -Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin | Arm 1P - Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin | Arm 2/Foll By Arm 1P-Low Dose Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin | Arm 2- Low Dose Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin | Arm 1P/Foll By Arm-1P/R-Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin
Started | 8 | 11 | 3 | 9 | 2
Completed | 7 | 11 | 3 | 9 | 2
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Not treated | 1 | 0 | 0 | 0 | 0
Period: Retreatment After First Drug Administrat
Arm/Group | Arm 1N -Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin | Arm 1P - Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin | Arm 2/Foll By Arm 1P-Low Dose Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin | Arm 2- Low Dose Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin | Arm 1P/Foll By Arm-1P/R-Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin
Started | 0 | 0 | 3 | 0 | 2
Completed | 0 | 0 | 3 | 0 | 2
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1N -Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin | Arm 1P - Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin | Arm 2/Foll By Arm 1P-Low Dose Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin | Arm 2- Low Dose Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin | Arm 1P/Foll By Arm-1P/R-Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin | Total
Number analyzed (Participants) | 8 | 11 | 3 | 9 | 2 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 10 | 3 | 9 | 2 | 32
  >=65 years | 0 | 1 | 0 | 0 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.28 (1.43) | 56.28 (13.39) | 31.07 (13.25) | 44.72 (3.66) | 53 (3.39) | 46.45 (13.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 4 | 1 | 11
  Male | 6 | 9 | 1 | 5 | 1 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 11 | 3 | 9 | 2 | 33
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 8 | 11 | 3 | 9 | 2 | 33
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 11 | 3 | 9 | 2 | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Grade 3-5 Adverse Events in Arm 1N and Arm 1P
Description: Number of participants with Grades 3-5 treatment-related adverse events were compared in Arm 1N and Arm 1P; and adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). Grade 3 is severe. Grade 4 is life-threatening, and Grade 5 is death related to adverse event.
Time Frame: 30 days after end of treatment
Population: One participant was not treated on Arm 1N. Pre-specified by the protocol, there are two combined reporting groups for this outcome. The first combined group (n=23) is all who received standard chemo (Arm 1N, Arm 1P, the retreatment of Arm 2/1P, and the initial treatment of Arm 1P/R). The second combined group (n=12) is all who received the reduced dose chemo (Arm 2, and the initial treatment of Arm 2/1P) This separates reporting of adverse events by the intensity of chemotherapy.
Measure: Count of Participants; unit: Participants
Groups:
- Grade 3 - Possibly Related Arm 1N, Arm 1P, Arm 2/1P, Arm 1/1P; Grade 3 - Probably Related Arm 1N, Arm 1P, Arm 2/1P, Arm 1/1P; Grade 3 - Definitely Related Arm 1N, Arm 1P, Arm 2/1P, Arm 1/1P: Grade 3 is severe.
  Cohort 1: 01 - Standard Chemo Prep Regimen. Young Tumor Infiltrating Lymphocytes (TIL) Plus High Dose Interleukin-2, Standard Chemo Preparative Regimen.
  Standard preparative regimen + Young Tumor Infiltrating Lymphocytes (TIL) Cells Aldesleukin: 720,000 IU/kg intravenous (IV) every eight hours (+/- 1 hour) beginning within 24 hours of cell infusion and continuing for up to 4 days (maximum 12 doses).
  Fludarabine: 25 mg/m^2/day intravenous piggy-back (IVPB) daily for 5 days Cyclophosphamide: 60 mg/kg/day X 2 days intravenous (IV) or 30 mg/kg/day X 2 days IV. Days -5 to -3 (low-dose arm-CLOSED): Cyclophosphamide 300 mg/m^2 IV over 60 minutes.
  Young TIL: Day 0: Cells will be infused intravenously (IV)
- Grade 4 - Possibly Related Arm 1N, Arm 1P, Arm 2/1P, Arm 1/1P; Grade 4 - Probably Related Arm 1N, Arm 1P, Arm 2/1P, Arm 1/1P; Grade 4 - Definitely Related Arm 1N, Arm 1P, Arm 2/1P, Arm 1/1P: Grade 4 is life-threatening.
  Cohort 1: 01 - Standard Chemo Prep Regimen. Young Tumor Infiltrating Lymphocytes (TIL) Plus High Dose Interleukin-2, Standard Chemo Preparative Regimen.
  Standard preparative regimen + Young Tumor Infiltrating Lymphocytes (TIL) Cells Aldesleukin: 720,000 IU/kg intravenous (IV) every eight hours (+/- 1 hour) beginning within 24 hours of cell infusion and continuing for up to 4 days (maximum 12 doses).
  Fludarabine: 25 mg/m^2/day intravenous piggy-back (IVPB) daily for 5 days Cyclophosphamide: 60 mg/kg/day X 2 days intravenous (IV) or 30 mg/kg/day X 2 days IV. Days -5 to -3 (low-dose arm-CLOSED): Cyclophosphamide 300 mg/m^2 IV over 60 minutes.
  Young TIL: Day 0: Cells will be infused intravenously (IV)
- Grade 5 - Possibly, Probably and/or Definitely Related Arm 1N, Arm 1P, Arm 2/1P, Arm 1/1P: Grade 5 is death related to adverse event.
  Cohort 1: 01 - Standard Chemo Prep Regimen. Young Tumor Infiltrating Lymphocytes (TIL) Plus High Dose Interleukin-2, Standard Chemo Preparative Regimen.
  Standard preparative regimen + Young Tumor Infiltrating Lymphocytes (TIL) Cells Aldesleukin: 720,000 IU/kg intravenous (IV) every eight hours (+/- 1 hour) beginning within 24 hours of cell infusion and continuing for up to 4 days (maximum 12 doses).
  Fludarabine: 25 mg/m^2/day intravenous piggy-back (IVPB) daily for 5 days Cyclophosphamide: 60 mg/kg/day X 2 days intravenous (IV) or 30 mg/kg/day X 2 days IV. Days -5 to -3 (low-dose arm-CLOSED): Cyclophosphamide 300 mg/m^2 IV over 60 minutes.
  Young TIL: Day 0: Cells will be infused intravenously (IV)
- Grade 3 - Possibly Related Arm 2, Arm 2/1P; Grade 3 - Probably Related Arm 2, Arm 2/1P; Grade 3 - Definitely Related Arm 2, Arm 2/1P: Grade 3 is severe.
  Cohort 1: 01 -> 01R - Standard Chemo Prep Regimen + Retreat. Young Tumor Infiltrating Lymphocytes (TIL) Plus High Dose Interleukin-2, Standard Chemo Preparative Regimen. 01R: Young Tumor Infiltrating Lymphocytes (TIL) Plus High Dose Interleukin-2, Standard Chemo (Retreat).
  Standard preparative regimen + Young Tumor Infiltrating Lymphocytes (TI) Cells + possible retreatment with standard preparative regimen + Young TIL Cells +pembrolizumab Aldesleukin: 720,000 IU/kg intravenous (IV) every eight hours (+/- 1 hour) beginning within 24 hours of cell infusion and continuing for up to 4 days (maximum 12 doses).
  Fludarabine: 25 mg/m^2/day intravenous piggy-back (IVPB) daily for 5 days Cyclophosphamide: 60 mg/kg/day X 2 days intravenous (IV) or 30 mg/kg/day X 2 days IV. Days -5 to -3 (low-dose arm-CLOSED): Cyclophosphamide 300 mg/m^2 IV over 60 minutes.
  Young TIL: Day 0: Cells will be infused intravenously (IV) Pembrolizumab: 2 mg/kg intravenous (IV) on Days -2, 21 (+/- 2 days), 42 (+/- 2 days), and 63 (+/- 2 days).
- Grade 4 - Possibly Related Arm 2, Arm 2/1P; Grade 4 - Probably Related Arm 2, Arm 2/1P; Grade 4 - Definitely Related Arm 2, Arm 2/1P: Grade 4 is life-threatening.
  Cohort 1: 01 -> 01R - Standard Chemo Prep Regimen + Retreat. Young Tumor Infiltrating Lymphocytes (TIL) Plus High Dose Interleukin-2, Standard Chemo Preparative Regimen. 01R: Young Tumor Infiltrating Lymphocytes (TIL) Plus High Dose Interleukin-2, Standard Chemo (Retreat).
  Standard preparative regimen + Young Tumor Infiltrating Lymphocytes (TI) Cells + possible retreatment with standard preparative regimen + Young TIL Cells +pembrolizumab Aldesleukin: 720,000 IU/kg intravenous (IV) every eight hours (+/- 1 hour) beginning within 24 hours of cell infusion and continuing for up to 4 days (maximum 12 doses).
  Fludarabine: 25 mg/m^2/day intravenous piggy-back (IVPB) daily for 5 days Cyclophosphamide: 60 mg/kg/day X 2 days intravenous (IV) or 30 mg/kg/day X 2 days IV. Days -5 to -3 (low-dose arm-CLOSED): Cyclophosphamide 300 mg/m^2 IV over 60 minutes.
  Young TIL: Day 0: Cells will be infused intravenously (IV) Pembrolizumab: 2 mg/kg intravenous (IV) on Days -2, 21 (+/- 2 days), 42 (+/- 2 days), and 63 (+/- 2 days).
- Grade 5 - Possibly, Probably and/or Definitely Related Arm 2, Arm 2/1P: Grade 5 is death related to adverse event.
  Cohort 1: 01 -> 01R - Standard Chemo Prep Regimen + Retreat. Young Tumor Infiltrating Lymphocytes (TIL) Plus High Dose Interleukin-2, Standard Chemo Preparative Regimen. 01R: Young Tumor Infiltrating Lymphocytes (TIL) Plus High Dose Interleukin-2, Standard Chemo (Retreat).
  Standard preparative regimen + Young Tumor Infiltrating Lymphocytes (TI) Cells + possible retreatment with standard preparative regimen + Young TIL Cells +pembrolizumab Aldesleukin: 720,000 IU/kg intravenous (IV) every eight hours (+/- 1 hour) beginning within 24 hours of cell infusion and continuing for up to 4 days (maximum 12 doses).
  Fludarabine: 25 mg/m^2/day intravenous piggy-back (IVPB) daily for 5 days Cyclophosphamide: 60 mg/kg/day X 2 days intravenous (IV) or 30 mg/kg/day X 2 days IV. Days -5 to -3 (low-dose arm-CLOSED): Cyclophosphamide 300 mg/m^2 IV over 60 minutes.
  Young TIL: Day 0: Cells will be infused intravenously (IV) Pembrolizumab: 2 mg/kg intravenous (IV) on Days -2, 21 (+/- 2 days), 42 (+/- 2 days), and 63 (+/- 2 days).
Arm/Group | Grade 3 - Possibly Related Arm 1N, Arm 1P, Arm 2/1P, Arm 1/1P | Grade 3 - Probably Related Arm 1N, Arm 1P, Arm 2/1P, Arm 1/1P | Grade 3 - Definitely Related Arm 1N, Arm 1P, Arm 2/1P, Arm 1/1P | Grade 4 - Possibly Related Arm 1N, Arm 1P, Arm 2/1P, Arm 1/1P | Grade 4 - Probably Related Arm 1N, Arm 1P, Arm 2/1P, Arm 1/1P | Grade 4 - Definitely Related Arm 1N, Arm 1P, Arm 2/1P, Arm 1/1P | Grade 5 - Possibly, Probably and/or Definitely Related Arm 1N, Arm 1P, Arm 2/1P, Arm 1/1P | Grade 3 - Possibly Related Arm 2, Arm 2/1P | Grade 3 - Probably Related Arm 2, Arm 2/1P | Grade 3 - Definitely Related Arm 2, Arm 2/1P | Grade 4 - Possibly Related Arm 2, Arm 2/1P | Grade 4 - Probably Related Arm 2, Arm 2/1P | Grade 4 - Definitely Related Arm 2, Arm 2/1P | Grade 5 - Possibly, Probably and/or Definitely Related Arm 2, Arm 2/1P
Number analyzed (Participants) | 23 | 23 | 23 | 23 | 23 | 23 | 23 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Participants
  ALT, SGPT (serum glutamic pyruvic transaminase) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  AST, SGOT(serum glutamic oxaloacetic transaminase) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Allergic reaction/hypersensitivity (including drug fever) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin (hyperbilirubinemia) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Confusion | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Diarrhea | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Febrile neutropenia | 0 | 3 | 4 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin | 4 | 2 | 6 | 1 | 0 | 0 | 0 | 2 | 1 | 3 | 0 | 0 | 0 | 0
  Hemorrhage, GU::Vagina | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypotension | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0
  Hypoxia | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Infection (documented clinically or microbiologically) w/Grade 3/4 neutrophils(ANC <1.0x10e9/L)Blood | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Left ventricular systolic dysfunction | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytes (total WBC) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphopenia | 0 | 0 | 1 | 0 | 2 | 14 | 0 | 0 | 0 | 0 | 0 | 2 | 9 | 0
  Nausea | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils/granulocytes (ANC/AGC) | 0 | 0 | 2 | 0 | 1 | 14 | 0 | 0 | 0 | 2 | 0 | 0 | 4 | 0
  PTT (Partial Thromboplastin Time) | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Phosphate, serum-low (hypophosphatemia) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets | 0 | 1 | 4 | 0 | 0 | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Renal failure | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Renal/Genitourinary - Other (Specify, oliguria) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Uric acid, serum-high (hyperuricemia) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Vomiting | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Weight loss | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Who Have a Clinical Response to Treatment (Objective Tumor Regression)
Description: Clinical response to treatment was assessed by the Response Evaluation Criteria In Solid Tumors (RECIST v1.0). Complete Response (CR) is disappearance of all target lesions. Partial Response (PR) is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD. Progressive Disease (PD) is at least a 20% increase in the sum of LD of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Stable Disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as references the smallest sum LD.
Time Frame: 4 weeks after cell infusion, then every 3 months x 3 and then every 6 months for 5 years, then per Principal Investigator (PI) discretion up to 5 years or disease progression
Population: The first combined group (n=16) is Arm 1P, the second treatment of Arm 2/1P, the initial treatment of Arm 1P/R. The second group (n=7) is Arm 1N (1/8 participants was not treated). The third group (n=12) is Arm 2 and the initial treatment of Arm 2/1P. The final group (n=2) will report the second treatment of Arm 1P/R. This enables reporting of the 37 treatments among the 32 treated participants separated by exposure to pembrolizumab/nivolumab and chemo dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1P - Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin | Arm 1N -Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin | Arm 2/Foll By Arm 1P-Low Dose Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin | Arm 1P/Foll By Arm-1P/R-Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin
Number analyzed (Participants) | 16 | 7 | 12 | 2
Participants
  First Treatment - Complete Response | 0 | 2 | 0 | NA — Participants in this group evaluated for second treatment only.
  First Treatment - Partial Response | 2 | 2 | 2 | NA — Participants in this group evaluated for second treatment only.
  First Treatment - Progressive Disease | 8 | 2 | 0 | NA — Participants in this group evaluated for second treatment only.
  First Treatment - Stable Disease | 3 | 1 | 1 | NA — Participants in this group evaluated for second treatment only.
  Second Treatment - Complete Response | 0 | NA — Participants in this group evaluated for first treatment only. | NA — Participants in this group evaluated for first treatment only. | 0
  Second Treatment - Partial Response | 1 | NA — Participants in this group evaluated for first treatment only. | NA — Participants in this group evaluated for first treatment only. | 1
  Second Treatment - Progressive Disease | 1 | NA — Participants in this group evaluated for first treatment only. | NA — Participants in this group evaluated for first treatment only. | 1
  Second Treatment - Stable Disease | 1 | NA — Participants in this group evaluated for first treatment only. | NA — Participants in this group evaluated for first treatment only. | 0

3. Primary Outcome: Overall Response Rate (ORR)
Description: Overall response is the best response recorded from the start of treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.0). Progression is at least a 20% increase in the sum of LD of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Date of cells until time of disease progression, up to approximately 67.2 months.
Population: Retreat Arm 1N and Arm 2 Foll By Arm 1P not treated.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1P - Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin | Arm 1N -Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin | Arm 2/Foll By Arm 1P-Low Dose Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin | Arm 1P/Foll By Arm-1P/R-Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin
Number analyzed (Participants) | 16 | 7 | 12 | 2
percentage of participants
  Initial Treatment: number analyzed (Participants) | 13 | 7 | 12 | 0
  Initial Treatment | 23.10 [8.2 to 50.3] | 57.10 [25 to 84.1] | 16.70 [3 to 44.8] |
  Retreat: number analyzed (Participants) | 3 | 0 | 0 | 2
  Retreat | 33.30 [1.7 to 88.2] |  |  | 50 [2.6 to 97.4]

4. Secondary Outcome: Number of Treatment-related Adverse Events for Participants Who Received Pembrolizumab
Description: Number of treatment-related adverse events for participants who received pembrolizumab. Adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v4.0.
Time Frame: Date treatment consent signed until approximately 4 weeks following last dose of Pembrolizumab, up to 4 weeks
Measure: Number; unit: Adverse events
Arm/Group | Arm 1P/Foll By Arm-1P/R-Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin
Number analyzed (Participants) | 2
Adverse events | 16

5. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time to disease progression following the start of treatment, and time to death following the start of treatment. Progression was assessed by the Response Evaluation Criteria In Solid Tumors (RECIST) v1.0 and is defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Date of cells until time of disease progression up to approximately 67.2 months.
Population: The first combined group (n=16) is Arm 1P, the second treatment of Arm 2/1P, the initial treatment of Arm 1P/R. The second group (n=7) is Arm 1N (1/8 participants was not treated). The third group (n=12) is Arm 2 and the initial treatment of Arm 2/1P. The final group (n=2) will report the second treatment of Arm 1P/R. This enables reporting of the 37 treatments among the 32 treated participants separated by exposure to pembrolizumab/nivolumab and chemo dose. 0 participants analyzed= not treated.
Measure: Median (Full Range); unit: Months
Arm/Group | Arm 1P - Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin | Arm 1N -Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin | Arm 2/Foll By Arm 1P-Low Dose Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin | Arm 1P/Foll By Arm-1P/R-Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin
Number analyzed (Participants) | 16 | 7 | 12 | 2
Months
  Initial Treatment: number analyzed (Participants) | 13 | 7 | 12 | 0
  Initial Treatment | 3.1 [1.3 to 14.6] | 7.9 [2 to NA] — Upper end was not reached because some participants had not progressed when taken off study. | 2.1 [0.9 to 12.8] |
  Retreat: number analyzed (Participants) | 3 | 0 | 0 | 2
  Retreat | 1.6 [0.1 to 5.3] |  |  | 32.5 [2.3 to NA] — Upper end was not reached because one participant had not progressed.

6. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from treatment start date until date of death, or date last known alive.
Time Frame: Date of cells until time to death, up until 90.1 months.
Population: As pre-specified by the protocol, participants will be reported by the initial treatment arm: Arm 1N (n=7; 1/8 participants were not treated), Arm 1P (n=13), Arm 2 (n=12).
Measure: Median (Full Range); unit: Months
Arm/Group | Arm 1P - Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin | Arm 1N -Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin | Arm 2- Low Dose Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin
Number analyzed (Participants) | 13 | 7 | 12
Months | 14.3 [2.3 to NA] — Insufficient number of participants with events. | NA [18.7 to NA] — Insufficient number of participants with events. | 15.1 [5.4 to NA] — Insufficient number of participants with events.

7. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from treatment start date until date of death, or date last known alive.
Time Frame: An average of 25.6 months.
Population: 1/8 participants were not treated in Arm 1N.
Measure: Median (Full Range); unit: Months
Groups:
- All Participants in Arms 1N, 1P, Arm 2/Foll By Arm 1P, Arm 2, and Arm 1P/Foll By Arm 1P/R: All Participants in Arms 1N, 1P, Arm 2/Foll By Arm 1P, Arm 2, and Arm 1P/Foll By Arm 1P/R.
Arm/Group | All Participants in Arms 1N, 1P, Arm 2/Foll By Arm 1P, Arm 2, and Arm 1P/Foll By Arm 1P/R
Number analyzed (Participants) | 32
Months | 17.5 [2.3 to NA] — Not applicable because some participants remain alive.

8. Secondary Outcome: Overall Progression Free Survival (PFS)
Description: as for outcome 5
Time Frame: Time to progression and time to death, approximately up to 67.2 months.
Population: 1/8 participants were not treated in Arm 1N.
Measure: Median (Full Range); unit: Months
Arm/Group | All Participants in Arms 1N, 1P, Arm 2/Foll By Arm 1P, Arm 2, and Arm 1P/Foll By Arm 1P/R
Number analyzed (Participants) | 32
Months | 3 [0.9 to NA] — Not applicable because some patients remain alive.

9. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 102 months and 9 days, 92 months and 19 days, 86 months and 9 days, 99 months and 16 days, and 86 months and 26 days for each group respectively.
Population: 1/8 participants were not treated on Arm 1N.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1N -Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin | Arm 1P - Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin | Arm 2/Foll By Arm 1P-Low Dose Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin | Arm 2- Low Dose Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin | Arm 1P/Foll By Arm-1P/R-Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin
Number analyzed (Participants) | 7 | 11 | 3 | 9 | 2
Participants | 7 | 9 | 3 | 9 | 2

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 102 months and 9 days, 92 months and 19 days, 86 months and 9 days, 99 months and 16 days, and 86 months and 26 days for each group respectively.
Description: 1/8 participants were not treated in Arm 1N.
Arm/Group | Arm 1N -Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin | Arm 1P - Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin | Arm 2/Foll By Arm 1P-Low Dose Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin | Arm 2- Low Dose Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin | Arm 1P/Foll By Arm-1P/R-Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin
All-Cause Mortality (participants affected / at risk) | 2/7 | 9/11 | 2/3 | 8/9 | 1/2
Serious Adverse Events (participants affected / at risk) | 3/7 | 6/11 | 1/3 | 2/9 | 1/2
Other Adverse Events (participants affected / at risk) | 7/7 | 9/11 | 3/3 | 9/9 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1N -Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin (N=7) | Arm 1P - Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin (N=11) | Arm 2/Foll By Arm 1P-Low Dose Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin (N=3) | Arm 2- Low Dose Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin (N=9) | Arm 1P/Foll By Arm-1P/R-Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin (N=2)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — (fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Hemoglobin (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Blood
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Platelets (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1N -Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin (N=7) | Arm 1P - Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin (N=11) | Arm 2/Foll By Arm 1P-Low Dose Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin (N=3) | Arm 2- Low Dose Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin (N=9) | Arm 1P/Foll By Arm-1P/R-Standard Chemotherapy Preparative Regimen + TIL + 720,000 IU/kg Aldesleukin (N=2)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bilirubin (hyperbilirubinemia) (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Creatinine (Investigations) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 0 (0) | 2 (2) | 2 (3) | 4 (4) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemoglobin (Investigations) | 2 (2) | 4 (6) | 3 (5) | 2 (2) | 1 (1)
Hemorrhage, GU::Vagina (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 2 (2) | 2 (3) | 4 (4) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Blood
Leukocytes (total WBC) (Investigations) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Investigations) | 4 (4) | 7 (10) | 2 (4) | 8 (8) | 2 (4)
Mood alteration::Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 4 (4) | 7 (7) | 2 (3) | 4 (4) | 2 (5)
PTT (Partial Thromboplastin Time) (Investigations) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Pain::Head/headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain::Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Platelets (Investigations) | 4 (4) | 6 (7) | 2 (2) | 0 (0) | 2 (5)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychosis (hallucinations/delusions) (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal/Genitourinary - Other (oliguria) (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rigors/chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular and nodal arrhythmia::Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision-blurred vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Leukocytes (total white blood cell (WBC) (Investigations) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Vision-blurred vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-15): https://cdn.clinicaltrials.gov/large-docs/19/NCT01993719/Prot_SAP_000.pdf
  • Informed Consent Form (2019-03-11): https://cdn.clinicaltrials.gov/large-docs/19/NCT01993719/ICF_001.pdf